CLINICAL TRIAL: NCT06877169
Title: Staged Kidney Transplantation During Combined Heart/Kidney Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Justin Steggerda, Assistant Professor of Surgery, Division of Abdominal Transplant Surgery, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003743
Record Dates: First submitted 2025-03-04; First posted 2025-03-14 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure; Chronic Kidney Disease; End-stage Kidney Disease
Keywords: combined heart and kidney transplant; simultaneous heart and kidney transplant; hypothermic oxygenated machine perfusion; organ preservation
MeSH Terms: conditions — Heart Failure; Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Delayed implantation with ex vivo machine perfusion of kidney allograft. (Experimental): Patients presenting for heart/kidney transplantation who consent to participate will be enrolled in this prospective, open-label, single-arm trial to undergo heart transplantation with planned delayed kidney transplantation with machine perfusion of the kidney allograft. Kidneys will be preserved using hypothermic oxygenated machine perfusion (HOPE) prior to transplantation. Timing of kidney implantation will be determined by recipient stability (e.g., vasopressor and inotrope requirements, coagulopathy, heart graft function) and allow for at least 6 hours of HOPE preservation. Both heart and kidney transplant procedures will follow standard of care techniques.
  Interventions: Other: Planned delayed implantation of kidney allograft with ex vivo machine perfusion kidney preservation.

INTERVENTIONS:
Other: Planned delayed implantation of kidney allograft with ex vivo machine perfusion kidney preservation. — During combined heart and kidney transplantation, heart and kidney allografts may be implanted during a single operative event, or with delayed kidney implantation in a second operative event. Timing of the delay is often determined by recipient stability and kidney availability; however, clinicians must balance recipient factors with accumulating cold ischemic time of the kidney allograft. This study uses hypothermic oxygenated machine perfusion to reduce ischemic injury to the kidney allograft and allow for improved recipient stability with planned delayed implantation of the kidney graft. Delays will allow for at least 6 hours of hypothermic oxygenated machine perfusion prior to implantation.

SUMMARY:
The primary purpose of this study is to evaluate the safety and efficacy of ex vivo machine perfusion with staged implantation of kidney allografts during combined heart/kidney transplantation.

DETAILED DESCRIPTION:
Combined heart and kidney transplantation (H/KTx) is the treatment of choice for patients with concomitant heart failure and chronic- or end-stage kidney disease. H/KTx presents a logistical challenge, often involving multiple surgical teams and requiring extended operative time to perform both heart and kidney transplants. Additionally, during heart transplantation, recipients require anticoagulation and multiple inotropes and vasopressors to support heart function early after implantation. While necessary, these may be detrimental to the newly implanted kidney allograft, potentially contributing to vasoconstriction, bleeding, hypotension, and worsening ischemia-reperfusion injury. Unfortunately, delaying implantation leads to extended cold ischemic time which also may be detrimental to the graft. Delayed graft function (DGF) of the kidney allograft is defined as the need for dialysis in the first seven days after transplantation and has been shown to be an important risk factor for graft loss following H/KTx. Ultimately, H/KTx requires balancing recipient stability with cold ischemic time to optimize kidney graft function. New perfusion technology adds oxygenation to the perfusate of the kidney allograft, thereby resuscitating the organ during preservation and reducing ischemia-reperfusion injury. This study seeks to evaluate the safety and efficacy of planned delayed implantation to allow for improved recipient stability and coagulopathy, while using hypothermic oxygenated machine perfusion (HOPE) for kidney preservation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or older) undergoing combined heart and kidney transplantation at Cedars-Sinai Medical Center.

Exclusion Criteria:

* Patients who undergo simultaneous heart/kidney transplantation in a single operative event due to medical necessity will be excluded.
* Patients with medical records flagged as "break-the-glass" or "research opt-out" within the center's electronic health record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2035-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of delayed graft function (DGF) of the kidney allograft | 7 days
  Delayed graft function (DGF) of the kidney allograft is defined as dialysis within the first 7 days post-transplant and will be monitored for all participants.
Number of patients with at least one adverse event | 90 days
  Safety endpoint will be assessed by monitoring for adverse events associated with either heart or kidney allografts within 90-days of initial operative event. Adverse events may include graft primary non-function, wound infection, urinary tract infection, ventilator-associated pneumonia, return to operating room, etc. Complications will be reported by Clavien-Dindo classification and analyzed as both those relating directly to the kidney transplant as well as overall incidence.

SECONDARY OUTCOMES:
Number of Patients with Heart Primary Graft Dysfunction | 24 hours
  Primary graft dysfunciton (PGD) of the heart allograft after transplant is defined as left ventricle, right ventricle, or biventricular dysfunction that occurs within 24 hours after surgery and is not associated with a discernible cause such as hyperacute rejection, pulmonary hypertension, massive blood product transfusion during surgery, or prolonged graft ischemic time. Grading will be done according to International Society of Heart and Lung Transplantation guidelines.
6 Month Kidney allograft function | 6 months
  Kidney function will be determined by estimated glomerular filtration rate at 6 months post-transplant.
12-month Kidney Allograft Function | 12 months
  Kidney function will be determined by estimated glomerular filtration rate at 12 months post-transplant.
intensive care unit length of stay | 1 year
  Patient intensive care unit length of stay following combined heart and kidney transplantation will be determined from date of transplant until date of transfer from intensive care unit to the patient ward.
Hospital Length of Stay | 1 year
  The duration of post-transplant hospital length of stay will be measured from day of transplant until day of discharge or death, up to 1 year post-transplant.
Number of readmissions | 90 days
  Patients will be assessed for number of readmissions following initial discharge during the first 90 days after combined heart and kidney transplantation.
Incidence of Kidney Allograft Rejection | 1 year
  Incidence of kidney rejection will be evaluated during the first post-transplant year. Rejection will be determined by biopsy findings and type of rejection (cell-mediated vs antibody mediated vs mixed) will be recorded.
Number of patients with Heart allograft rejection | 1 year
  Incidence of heart rejection will be evaluated during the first post-transplant year. Rejection will be determined by biopsy findings and type of rejection (cell-mediated vs antibody mediated vs mixed) will be recorded.
36-month kidney allograft function | 36 months
  Long-term graft function and survival will be assessed by estimated glomerular filtration rate (eGFR) at 3-years post-transplant. Graft loss before 3-years will be determined by death or return to dialysis and will be recorded in lieu of graft function.

CONTACTS AND LOCATIONS:
Overall Officials: Justin A Steggerda, M.D., Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kobashigawa J, Zuckermann A, Macdonald P, Leprince P, Esmailian F, Luu M, Mancini D, Patel J, Razi R, Reichenspurner H, Russell S, Segovia J, Smedira N, Stehlik J, Wagner F; Consensus Conference participants. Report from a consensus conference on primary graft dysfunction after cardiac transplantation. J Heart Lung Transplant. 2014 Apr;33(4):327-40. doi: 10.1016/j.healun.2014.02.027. Epub 2014 Mar 5. PMID 24661451
- [Background] Jochmans I, Brat A, Davies L, Hofker HS, van de Leemkolk FEM, Leuvenink HGD, Knight SR, Pirenne J, Ploeg RJ; COMPARE Trial Collaboration and Consortium for Organ Preservation in Europe (COPE). Oxygenated versus standard cold perfusion preservation in kidney transplantation (COMPARE): a randomised, double-blind, paired, phase 3 trial. Lancet. 2020 Nov 21;396(10263):1653-1662. doi: 10.1016/S0140-6736(20)32411-9. PMID 33220737
- [Background] Lutz AJ, Nagaraju S, Sharfuddin AA, Garcia JP, Saleem K, Mangus RS, Goggins WC. Simultaneous Heart-kidney Transplant With Planned Delayed Implantation of the Kidney Graft After Ex Vivo Perfusion. Transplantation. 2023 Sep 1;107(9):2043-2046. doi: 10.1097/TP.0000000000004661. Epub 2023 Jun 5. PMID 37271866
- [Background] Ruzza A, Czer LS, Trento A, Esmailian F. Combined heart and kidney transplantation: what is the appropriate surgical sequence? Interact Cardiovasc Thorac Surg. 2013 Aug;17(2):416-8. doi: 10.1093/icvts/ivt172. Epub 2013 Apr 24. PMID 23615433